CLINICAL TRIAL: NCT07050095
Title: Randomized Clinical Trial for Comparison Between the Anxiolytic Effect of Virtual Reality Immersion Versus Midazolam Premedication in Patients Undergoing Dacryocystorhinostomy Surgery
Brief Title: Anxiolytic Effect of Virtual Reality Immersion Versus Midazolam Premedication in Patients Undergoing Dacryocystorhinostomy Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hebatallah Salah Abdelhamid, Lecturer of Anesthesia, Surgical Critical Care and Pain Management Department, Faculty of Medicine, Cairo University, Cairo, Egypt., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MS-526-2023
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Anxiolytic Effect; Virtual Reality Immersion; Midazolam; Premedication; Dacryocystorhinostomy
MeSH Terms: interventions — Midazolam

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality Group (Experimental): Patient will undergo virtual reality (VR) immersion using oculus.
  Interventions: Other: Virtual Reality Group
- Midazolam Group (Active Comparator): Patient will receive midazolam premedication only.
  Interventions: Drug: Midazolam Group

INTERVENTIONS:
Other: Virtual Reality Group — Patient will undergo virtual reality (VR) immersion using oculus.
  Other Names: Guided Meditation VR
  Arms: Virtual Reality Group
Drug: Midazolam Group — Patient will receive midazolam premedication only.
  Other Names: Midazolam
  Arms: Midazolam Group

SUMMARY:
The aim is to investigate the anxiolytic effect, and hemodynamic stability of using virtual reality immersion in adult patients undergoing Dacryocystorhinostomy (DCR) operation under general anesthesia and to compare its effect to that of using Midazolam as a premedication.

DETAILED DESCRIPTION:
Anxiety is a negative emotion characterized by fear, tension, and nervousness. Preoperative anxiety is anxiety due to disease, hospitalization, or scheduled surgery. The most common causes of preoperative anxiety are waiting for surgery, worrying about the operation outcome, being separated from family, anticipating postoperative pain, losing independence, and being afraid of surgery, pain, and death.

Midazolam reduces anxiety by acting on GABAA receptors, resulting in sedation; however, the benefit of midazolam premedication remains debatable, and the drug's side effects include paradoxical reactions, oversedation, reduced blood pressure, and respiratory depression. Regarding this, some clinicians challenge the clinical benefits of benzodiazepine premedication and contend that non-pharmacological treatments alone are sufficient to minimize preoperative anxiety.

Virtual reality is a computer technology that creates the sensation of being immersed in a simulated three-dimensional environment in which the user can interact with the virtual environment. It has also been suggested as a non-pharmaceutical alternative for lowering surgical pain and anxiety.

Dacryocystorhinostomy (DCR) is a procedure that circumvents the blocked tear duct and offers an alternate path for the drainage of tears from the eye to the nose and is most effectively performed under a general anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65.
* Both sexes.
* American Society of Anesthesiologists (ASA) classification: I - II.
* Patient undergoing Dacryocystorhinostomy Surgery (DCR) operation under general anesthesia.

Exclusion Criteria:

* Patient refusal.
* Patients with cardiac diseases.
* Patients with renal diseases.
* Patients with drug sensitivity and seizures.
* Substance abuse and addiction.
* Claustrophobia.
* Patients with cerebrovascular disease.
* Psychiatric and cognitive disorder.
* Patients with severe teary eyes and blurring of vision.
* Patients who express discomfort during the test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Anxiety Score | 15-minute after intervention
  Beck Anxiety Inventory (BAI) score change measured from pre- to post-intervention (virtual reality (VR) or midazolam). The score ranges from 0 to 63. A greater reduction indicates better anxiolytic effect.5 minutes before intervention and Immediately after the 15-minute virtual reality (VR) session or midazolam injection

SECONDARY OUTCOMES:
Heart rate (HR) | After intubation (Up to 2 hours)
  Heart rate (HR) measured to assess perioperative hemodynamic response to anxiolytic intervention.At four time points: T1 (initial on the day of surgery), T2 (before induction), T3 (before intubation), and T4 (after intubation).
Systolic blood pressure (SBP) | After intubation (Up to 2 hours)
  Systolic blood pressure (SBP) recorded to evaluate cardiovascular response to premedication and induction.At four time points: T1 (initial on the day of surgery), T2 (before induction), T3 (before intubation), and T4 (after intubation).
Diastolic blood pressure (DBP) | After intubation (Up to 2 hours)
  Diastolic blood pressure (DBP) measured to monitor hemodynamic changes related to stress and sedation.At four time points: T1 (initial on the day of surgery), T2 (before induction), T3 (before intubation), and T4 (after intubation).
Mean blood pressure (MBP) | After intubation (Up to 2 hours)
  Mean blood pressure (MBP) recorded to reflect overall perfusion pressure during perioperative period.At four time points: T1 (initial on the day of surgery), T2 (before induction), T3 (before intubation), and T4 (after intubation).
Patient Satisfaction | 2 hours Post intervention
  Survey with options: very satisfied, satisfied, undecided, or unsatisfied
Incidence of Complications | First 30 minutes post-extubation
  Presence of headache, dizziness, nausea, or virtual reality (VR)related discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author